CLINICAL TRIAL: NCT02797808
Title: Effects of Sertraline on Brain Connectivity in Adolescents With OCD (Obsessive-Compulsive Disorder)
Brief Title: Effects of Sertraline on Brain Connectivity in Adolescents With OCD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1105M99532; 5R21MH101395-02 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: OCD
Keywords: OCD
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Children with OCD (Experimental): Children with obsessive compulsive disorder, not currently on medication for OCD
  Interventions: Drug: Sertraline
- Healthy Control Children (Active Comparator): Children without obsessive compulsive disorder
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Sertraline — Impact of sertraline on functional brain connectivity
  Other Names: Zoloft
  Arms: Children with OCD
Other: No Intervention — Healthy control non-intervention
  Arms: Healthy Control Children

SUMMARY:
The investigators will examine how treatment with sertraline for 12 weeks impacts frontal-striatal-thalamic circuitry (FSTC) in this OCD sample.

DETAILED DESCRIPTION:
To examine FSTC using advanced multi-modal imaging techniques, including resting-state functional magnetic resonance imaging (R-fMRI) and high angular resolution diffusion imaging (HARDI), in 25 medication-free adolescents youths with OCD (ages 8-17) in comparison with 25 matched healthy controls.

Hypotheses: (A) Based on the pilot data, adolescents youths with OCD will show lower functional connectivity in FSTC at baseline when compared with controls, and , lower functional connectivity in FSTC will correlate with greater severity on CY-BOCS. (B) Adolescents Youths with OCD will also show abnormalities in structural connectivity in FSTC at baseline when compared with controls, and structural and functional connectivity will be related. (C) The investigators will explore relations between OCD dimensions and functional connectivity measures, and predict that the repeating/ordering dimension will correlate with orbitofrontal cortex (OFC) connections, hoarding will correlate with rostral anterior cingulate cortex (ACC) connections, and forbidden thoughts will correlate with caudal ACC connections.

To investigate how sertraline impacts functional connectivity in FSTC in adolescents with OCD.

Hypothesis: After 12 weeks of sertraline treatment, functional connectivity measures within FSTC for the OCD group will (on average) increase compared to baseline and will no longer be significantly different when compared with controls. Non-responders may show a different pattern (i.e. failure to show these changes).

ELIGIBILITY:
Inclusion Criteria (OCD):

* OCD as the primary Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnosis based on the Anxiety Disorders Interview Schedule (ADIS) for DSM-IV, Child Version
* Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) score of greater than 15

Exclusion Criteria (OCD):

* lifetime diagnosis of bipolar disorder, schizophrenia, or substance abuse/dependence on ADIS
* Intelligence Quotient (IQ) < 80 on Wechsler Abbreviated Scales of Intelligence (WASI)
* positive urine drug screen
* MRI-incompatible features (e.g., metal implants, claustrophobia)
* current or recent trial of psychotropic medication (within the past 4 8 weeks or past 6 12 weeks for fluoxetine)
* non-response in > 2 selective serotonin reuptake inhibitor (SSRI) trials of adequate dose/duration
* positive pregnancy test
* history of seizure disorder or serious head injury

Inclusion Criteria (Controls):

* Healthy 8-17 year olds

Exclusion criteria (controls):

* No psychiatric diagnoses
* No immediate family history of OCD

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2013-08; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail A Bernstein, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernstein GA, Mueller BA, Schreiner MW, Campbell SM, Regan EK, Nelson PM, Houri AK, Lee SS, Zagoloff AD, Lim KO, Yacoub ES, Cullen KR. Abnormal striatal resting-state functional connectivity in adolescents with obsessive-compulsive disorder. Psychiatry Res Neuroimaging. 2016 Jan 30;247:49-56. doi: 10.1016/j.pscychresns.2015.11.002. Epub 2015 Nov 19. PMID 26674413
- [Derived] Bernstein GA, Cullen KR, Harris EC, Conelea CA, Zagoloff AD, Carstedt PA, Lee SS, Mueller BA. Sertraline Effects on Striatal Resting-State Functional Connectivity in Youth With Obsessive-Compulsive Disorder: A Pilot Study. J Am Acad Child Adolesc Psychiatry. 2019 May;58(5):486-495. doi: 10.1016/j.jaac.2018.07.897. Epub 2018 Oct 30. PMID 30768407

RESULTS

PARTICIPANT FLOW:
Groups:
- Obsessive-compulsive Disorder: Sertraline: Impact of sertraline on functional brain connectivity
- Healthy Controls: No Intervention: Healthy control non-intervention
Period: Overall Study
Arm/Group | Obsessive-compulsive Disorder | Healthy Controls
Started | 23 | 18
Completed | 16 | 15
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obsessive-compulsive Disorder | Healthy Controls | Total
Number analyzed (Participants) | 23 | 18 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 18 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.6) | 13.4 (2.9) | 13.4 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 13 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 4 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 18 | 41
CY-BOCS Total Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) a clinician-rated semi-structured instrument assessing OCD severity over the previous 7 days in children ages 6 to 17 years. Items are scored from 0 (none) to 4 (extreme) and total score ranges from 0 to 40 with higher scores indicating greater impairment. All 19 items are rated, but only items 1-10 are used to determine the total score. The total CY-BOCS score is the sum of items 1-10.
  units on a scale | 24.8 (6.9) | 0 (0) | 24.8 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: CY-BOCS Total Score at 12-weeks
Description: The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) a clinician-rated semi-structured instrument assessing OCD severity over the previous 7 days in children ages 6 to 17 years. Items are scored from 0 (none) to 4 (extreme) and total score ranges from 0 to 40 with higher scores indicating greater impairment. All 19 items are rated, but only items 1-10 are used to determine the total score. The total CY-BOCS score is the sum of items 1-10; the obsession and compulsion subtotals are the sums of items 1-5 and 6-10, respectively. At this time, items 1A and 6A are not being used in the scoring. Items 17 (global severity) and 18 (global improvement) are adapted from the Clinical Global Impression Scale to provide measures of overall functional impairment associated with the presence of obsessive-compulsive symptoms.
Time Frame: 12 weeks
Population: 2 additional participants with OCD and 1 Healthy Control were removed from this analysis due to motion effects in the neuroimaging data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children With OCD | Healthy Control Children
Number analyzed (Participants) | 14 | 14
units on a scale | 14.1 (8.5) | 0 (0)

2. Primary Outcome: Longitudinal 2-Group Resting State Functional Conectivity (RSFC) Analyses
Description: Participants had whole brain fMRI at baseline &12 weeks. Whole brain connectivity in 6 striatal ROIs was performed. Two-way mixed effects ANOVAs were performed with FEAT. Clusters were significant if p <.0042 based on .05/(6 ROIs x 2 tests/ROI). Mean z-score was found for each time point in each subject's connectivity map in each significant cluster. Within-group paired-sample t tests examined RSFC change over time in these metrics for each group. To investigate group X time interactions from the 2-way ANOVA, we compared mean z-scores within each significant cluster at baseline & 12 weeks. Resulting numbers represented striatal connectivity for each individual at each time point. Within group paired sample t-tests examined RSFC change over time for each group. Bonferroni correction was applied to alpha level (2-tailed, p<0.5/6 =.0083) for multiple testing. We do not have an a priori hypothesis as to whether increase or decrease in RSFC is a better outcome. Unit of measure is z-score.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Children With OCD | Healthy Control Children
Number analyzed (Participants) | 14 | 14
z score
  Connectivity z-scores for right putamen at baseline | 0.15 (1.04) | 1.44 (1.06)
  Connectivity z-scores for right putamen at 12 weeks | 1.89 (0.85) | 0.60 (0.98)
  Connectivity z-scores for left putamen at baseline | 1.46 (1.14) | 2.41 (1.19)
  Connectivity z-scores for left putamen at week 12 | 3.03 (1.54) | 0.89 (0.99)
Statistical Analysis 1: Comparison: Children With OCD vs Healthy Control Children; Test type: Superiority; p < 0.0083, ANOVA — Independent-sample t tests were used to compare the RSFC metrics between groups at baseline and 12 weeks. Bonferroni correction was applied to the alpha level (2-tailed, p<.05/6= .0083) for multiple testing

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Obsessive-compulsive Disorder | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/18
Other Adverse Events (participants affected / at risk) | 8/23 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obsessive-compulsive Disorder (N=23) | Healthy Controls (N=18)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obsessive-compulsive Disorder (N=23) | Healthy Controls (N=18)
Medication Side Effect (General disorders) | 8 (21) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02797808/Prot_SAP_000.pdf